CLINICAL TRIAL: NCT03765008
Title: The Effect of Water Intake on Glucose Regulation: A Pilot Study
Brief Title: The Effect of Water Intake on Glucose Regulation
Acronym: INDIGO-I
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not get funded
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Stavros Kavouras, Professor of Nutrition, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FP00018531
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Glucose Metabolism Disorders; Dehydration (Physiology); Water Deprivation
Keywords: water; vasopressin
MeSH Terms: conditions — Glucose Metabolism Disorders; Dehydration; Diabetes Insipidus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Water intake (Active Comparator): 5-days of High water intake according to IOM guidelines
  Interventions: Other: Water intake manipulation
- Low Water Intake (Experimental): 5-days of Low water intake of 500 mL/day
  Interventions: Other: Water intake manipulation

INTERVENTIONS:
Other: Water intake manipulation — for 5 days prior to each experiment subjects will undergo manipulation of their water intake.

SUMMARY:
There is a growing body of evidence suggesting low water intake and elevated levels of the hormone vasopressin exacerbate glucose regulation. This project will examine the physiological mechanism by which low water intake impairs glucose homeostasis.

In the current proposal we aim to: 1) quantify the degree of glucose impairment as a response to elevated vasopressin due to low water intake and 2) identify the physiological mechanism by which elevated vasopressin, as a response to low water intake, impairs glucose regulation

ELIGIBILITY:
Inclusion Criteria:

BMI 27.5-35

Exclusion Criteria:

* BMI <27.5 or >35
* high physical activity
* diabetes
* impaired liver or kidney function
* cardiovascular disease
* weight change of more than 3 kg in the past month
* pregnancy
* previous surgery on digestive tract (except appendectomy)
* fluid balance will be exclusionary such as
* serotonin re-uptake inhibitors.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-11 (Estimated); Primary Completion 2019-04-03 (Estimated); Study Completion 2019-04-29 (Estimated)

PRIMARY OUTCOMES:
amount of glucose metabolized M | 220-240 min & 340-360 min of the protocol
  amount of glucose metabolized during the euglycemic & Hyperglycemic clamp
metabolic clearance rate for insulin | 220-240 min & 340-360 min of the protocol
  metabolic clearance rate for insulin during the euglycemic & Hyperglycemic clamp
quantity of glucose metabolized per unit plasma insulin concentration | 220-240 min & 340-360 min of the protocol
  quantity of glucose metabolized per unit plasma insulin concentration during the euglycemic & Hyperglycemic clamp
Rate of glucose appearance & disappearance | 220-240 min & 340-360 min of the protocol
  Rate of glucose appearance & disappearance during the euglycemic & Hyperglycemic clamp

SECONDARY OUTCOMES:
Plasma copeptin | 0 min, 240 min & 360 min of the protocol
  Plasma copeptin in response to water manipulation
glucagon | 0 min, 240 min & 360 min of the protocol
  glucagon in response to water manipulation
Cortisol | 0 min, 240 min & 360 min of the protocol
  Cortisol in response to water manipulation

IPD SHARING:
Plan to Share IPD: No